## ORI IRB# 00000278

Protocol Version 8/19/2020

Official Title: Talk STEM Familia: Dual-Language Academic Vocabulary-Building Technology to

Improve Educational, Career, and Health Outcomes Among Latinx Students

Principal Investigators: Jessie Marquez and Patricia Vadasy, Ph.D.

Oregon Research Behavior Interventions Strategies, dba Influents Innovations

Award No. 2 R44 MD013619-02

Final Version Dated: 5/30/2023

## Parental Informed Consent for Talk STEM Familia Evaluation Study

You and your 4<sup>th</sup>-8<sup>th</sup> grade child are invited to participate in a research study to test Talk STEM Familia, a Spanish/English Alexa skill (app) with lessons and practice games in the vocabulary words that support success in STEM (science, technology, engineering, and math).

There are growing opportunities in STEM fields. Using STEM words at home in Spanish and English prepares students for success.

The project is led by *Jessie Marquez and Patricia Vadasy*, *Ph.D.* of Influents Innovations in Eugene, OR.

The Talk STEM study is funded by the National Institute of Minority Health Disparities (grant # 2 R44 MD013619-02).

After reviewing the study details, please ask any questions you might have before agreeing to participate.

## If You Decide to Participate, You will be Asked to:

- Be randomly selected (by chance) to use the Talk STEM Familia technology in the first half of the study period or the second half.
- Complete an online survey on demographics, vocabulary, and how confident you feel helping your child with academic subjects.
- Provide permission for your child to fill out an online survey about vocabulary and how confident he/she feels about academic subjects.
- Receive an Alexa Echo Dot by mail.
- If you are randomly selected to be in the first group, receive links to videos about how to set up the Echo Dot and use the Talk STEM Familia skill. We will check in with you to see if you need any help with this.
- We will provide you with an Amazon account so you can access the Talk STEM Familia skill on your Alexa Echo Dot.
- Then, for 6 months, you will receive reminder text messages to use Talk STEM Familia with your child 3/days a week for approximately 10-minutes, at your convenience.
- After 3 months, all participants (parents/students) will complete a 2<sup>nd</sup> survey on vocabulary and confidence using vocabulary. Participants in the first group will also receive a survey about how useful and engaging Talk STEM is, and how well it meets your family needs.
- At that point, you and your child will receive \$100 in the form of check or gift card, whichever you prefer.
- Finally, at the end of the 6 months, all participants (parent/students) will complete a 3<sup>nd</sup> survey on vocabulary and confidence using vocabulary. Participants in the first group will also complete a survey about how useful and engaging Talk STEM is, and how well it meets your family needs.
- At this time, you and your child will receive a final \$100 in the form of check or gift card, whichever you prefer.
- At this time, we will also close the Amazon accounts of participants in the first group and

- participants will then be able to set up or use their own Amazon account.
- If you were randomly slected to be in the second group, you will be given access to the Talk STEM Familia technology.

### Risks and What Will Be Done to Reduce the Risks

Here are some risks involved for you and your child as participants:

- 1. We collect and store names, email addresses, mailing addresses, and phone numbers to communicate with you about the study. Because it is possible that someone who is not authorized could see it, we take these precautions to protect your confidentiality and your information:
  - a. Any information you or your child give us will be kept strictly confidential. We will keep all information in a locked file. We will remove all names from all the information we get from you (except this consent form). An ID # will be assigned to the information you give us, and only authorized staff will have access to the locked file that links your name to your ID#.
  - b. The Amazon account we set up for you will not have your name on it. We will use a number instead.
  - c. We have a Certificate of Confidentiality, a legal assurance from the federal government that will help us protect your privacy even if the records are subpoenaed. We will not give information to anyone unless you provide a signed release telling us to do so, or unless we have reason to suspect: 1) abuse, neglect, or endangerment of a child or elder; 2) or that anyone is in immediate danger of seriously hurting himself/herself or someone else. In these situations, we may have to make a report to the appropriate authorities.
  - d. If the U. S. Department of Health and Human Services (DHHS) audits our research project, they can have access to information about you. However, they cannot report it to the police or use it for any reason besides the audit.
  - e. A description of this clinical trial will be available on <a href="http://www.ClinicalTrials.gov">http://www.ClinicalTrials.gov</a>. This website will not include information that can identify you. At most, the website will include a summary of the research results. At the very end of the project, we will post a study consent form to the same website. The consent form will not have names on it. You can search this website at any time.
  - f. The information that you give us will be used only for this study. We will not share information about you with others or use it in future studies without your consent. There is still a chance that someone could figure out that the information is about you.
- 2. You may have questions or concerns about smart speakers like the Echo Dot and your privacy.
  - a. We will show you the lights on the Echo Dot that indicate when it captures and sends audio to the cloud-based system. We will show you how the voice system works and how to disable the microphone so that no audio/sound can be captured and sent to the cloud. You will also be able to keep the Echo Dot unplugged between use.
  - b. Unidentifiable usage data is kept by Amazon to improve the quality of their speech

recognition programs. Other usage data is stored in the password protected account of the user. In this study, the research project staff will manage and own the accounts and will have access to usage data within the account. Since the account will be unidentifiable, research staff will not be able to link this usage data to specific families. We will keep unidentifiable usage data in the research project's database. This will include data such as time spent using the skill, percentage correct, progress, and how often a word was practiced.

3. You and/or your child might feel uncomfortable if you are unsure about how to answer questions on the surveys. You will be able to call or text us and we will provide support.

# Benefits to You and Your Child for Participation

You and your child could enjoy learning new vocabulary words and using them to talk about school and home interests. You and your child could enjoy being a part of research that supports the educational and health outcomes of others.

## Your Right to Withdraw from the Study

Your participation is completely voluntary and private. While your child's school has shared this research opportunity with you, no one at your child's school will know who chooses to participate or not. If you decide not to participate it will not affect your child at school. If you decide to participate, you can stop participating at any time without penalty.

## **Request for more information**

If you have questions about the research at any time, or if you have a visual or other impairment and require this material in another format, please call: Natasha Compton, Research Assistant (541) 484-2123 x2994 1776 Millrace Dr., Eugene, OR 97403. ORI's TDD number is 800-735-2900

If you have questions about your rights as a research subject, call the Office for the Protection of Human Subjects, Oregon Research Institute, (541) 484-2123. ORI's TDD number is 800-735-2900.

Do you have any questions?

We have sent you a copy of this form to keep. Saying that you do want to participate in this study indicates that you:

- (1) understand the information provided today,
- (2) agree to participate,
- (3) consent to your child's participation,
- (4) may withdraw your consent at any time and stop participating at any time without penalty,
- (5) may withdraw your consent for your child's participation at any time without penalty to you or your child
- (6) have received a copy of this consent form.
- ¿Do you want to participate in this study? Sí No
- ¿Do you allow your child to participate in this study? Sí No

| Printed Name (of parent): |
|---|
| Child's First Name: |
| Date: |
| CHILD AGREEMENT TO PARTICIPATE |
| Evaluation Study |
| We are inviting you and your family to participate in a study to test the Mi Familia STEM app and smart speaker technology. Mi Familia STEM is a Spanish/English word learning game for smartphones and smart speakers. It includes words like: <i>evidence, variable, dimension, and hypothesis</i> and other words that help students in school. |
| If you decide to participate, we'll ask you to use Mi Familia STEM for about 10-minutes, 3 times/week, for 6 months. |
| We'll also ask you to complete some online surveys. |
| You and your parent will receive a smart speaker to keep and \$200. |
| Your parents have already told us that it is okay for you to participate if you want to. You don't have to participate if you don't want to. |
| If you decide you <b>do</b> want to participate now, you can change your mind at any time. |
| Do you have questions? |
| Would you like to participate in the study? Yes No |
| Student Name: |

# Consentimiento Informado para Padres para Estudio de Evaluación de Mi Familia STEM (Talk STEM II)

Usted y su hijo/a de cuarto a octavo grado están invitados a participar en un estudio de investigación para probar Mi Familia STEM, una aplicación y una habilidad (aplicación) de

Date: \_\_\_\_\_

Alexa en español/inglés con lecciones y juegos de práctica en las palabras del vocabulario que respaldan el éxito en STEM (ciencia, tecnología, ingeniería y matemáticas).

Cada vez hay más oportunidades en los campos de STEM. El uso de palabras STEM en casa en español e inglés prepara a los estudiantes para el éxito.

El proyecto está dirigido por *Jessie Marquez y Patricia Vadasy, Ph.D.* de Influents Innovations en Eugene, Oregón.

El estudio Talk STEM está financiado por el Instituto Nacional de Disparidades de Salud de las Minorías (subvención # 2 R44 MD013619-02).

Después de revisar los detalles del estudio, haga cualquier pregunta que pueda tener antes de aceptar participar.

## Si decide participar:

- Será seleccionado al azar (por casualidad) para usar la tecnología Mi Familia STEM en la primera mitad del período de estudio o la segunda mitad.
- Completará una encuesta en línea sobre demografía, vocabulario y de qué tan seguro se siente al ayudar a su hijo/a con las materias académicas.
- Permitirá que su hijo/a complete una encuesta en línea sobre vocabulario y de qué tan seguro/a se siente acerca de las materias académicas.
- Recibirá un Alexa Echo Dot por correo.
- Si es seleccionado/a al azar para estar en el primer grupo, recibirá enlaces a videos sobre cómo configurar el Echo Dot y usar la habilidad Mi Familia STEM. Nos comunicaremos con usted para ver si necesita ayuda.
- Le proporcionaremos una cuenta de Amazon para que pueda acceder a la habilidad Mi Familia STEM en su Alexa Echo Dot.
- Luego, durante 6 meses, recibirá mensajes de texto recordatorios para usar Mi Familia STEM con su hijo/a 3 veces a la semana durante aproximadamente 10 minutos, según su conveniencia.
- Después de 3 meses, todos los participantes (padres/estudiantes) completarán una segunda encuesta sobre vocabulario y confianza usando dicho vocabulario.
- En ese momento, usted y su hijo/a recibirán \$100 en forma de cheque o tarjeta de regalo, lo que prefieran.
- Finalmente, al final de los 6 meses, todos los participantes (padres/estudiantes) completarán una tercera encuesta sobre vocabulario y confianza usando dicho vocabulario. Los participantes del primer grupo también completarán una encuesta sobre lo útil y atractivo que es Talk STEM, y qué tan bien satisface las necesidades de su familia.
- En ese momento, usted y su hijo/a recibirán la última suma de \$100 en forma de cheque o tarjeta de regalo, lo que prefieran.
- En ese momento, también cerraremos las cuentas de Amazon de los participantes del primer grupo y los participantes podrán configurar o usar su propia cuenta de Amazon.

• Si fue seleccionado al azar para estar en el segundo grupo, se le dará acceso a la tecnología Mi Familia STEM.

## Riesgos y Qué Se Hará para Reducir los Riesgos

Estos son algunos de los riesgos involucrados para usted y su hijo/a como participantes:

- 1. Recopilamos y almacenamos nombres, direcciones de correo electrónico, direcciones postales y números de teléfono para comunicarnos con usted sobre el estudio. Debido a que es posible que alguien no autorizado pueda verlo, tomamos estas precauciones para proteger su confidencialidad y su información:
  - a. Cualquier información que usted o su hijo/a nos proporcione se mantendrá estrictamente confidencial. Mantendremos toda la información en un archivo bloqueado. Eliminaremos todos los nombres de toda la información que obtengamos de usted (excepto este formulario de consentimiento). Se asignará un número de identificación a la información que nos proporcione, y solo el personal autorizado tendrá acceso al archivo bloqueado que vincula su nombre con su número de identificación.
  - b. La cuenta de Amazon que configuramos para usted no tendrá su nombre. En su lugar, usaremos un número.
  - c. Tenemos un Certificado de Confidencialidad, una garantía legal del gobierno federal que nos ayudará a proteger su privacidad incluso si los registros son citados. No proporcionaremos información a nadie a menos que usted proporcione una autorización firmada que nos indique que lo hagamos, o a menos que tengamos motivos para sospechar: 1) abuso, negligencia o puesta en peligro a un niño o anciano; 2) o que alguien esté en peligro inmediato de lastimarse gravemente a sí mismo o a otra persona. En estas situaciones, es posible que tengamos que informar a las autoridades correspondientes.
  - d. Si el Departamento de Salud y Servicios Humanos de los EE. UU. (DHHS) audita nuestro proyecto de investigación, pueden tener acceso a información sobre usted. Sin embargo, no pueden denunciarlo a la policía ni utilizarlo por ningún motivo además de la auditoría.
  - e. Una descripción de este ensayo clínico estará disponible en http://www.ClinicalTrials.gov. Este sitio web no incluirá información que pueda identificarlo. Como máximo, el sitio web incluirá un resumen de los resultados de la investigación. Al final del proyecto, publicaremos un formulario de consentimiento para el estudio en el mismo sitio web. El formulario de consentimiento no tendrá nombres. Puede buscar en este sitio web en cualquier momento.
  - f. La información que nos proporcione se utilizará únicamente para este estudio. No compartiremos información sobre usted con otros ni la usaremos en estudios futuros sin su consentimiento. Todavía existe la posibilidad de que alguien se dé cuenta de que la información es sobre usted.
- 2. Es posible que tenga preguntas o inquietudes sobre los altavoces inteligentes como el Echo Dot y su privacidad.

- a. Le mostraremos las luces del Echo Dot que indican cuándo captura y envía audio al sistema basado en la nube. Le mostraremos cómo funciona el sistema de voz y cómo deshabilitar el micrófono para que no se pueda capturar ni enviar audio/sonido a la nube. También podrá mantener el Echo Dot desenchufado entre usos.
- b. Amazon conserva los datos de uso no identificables para mejorar la calidad de sus programas de reconocimiento de voz. Otros datos de uso se almacenan en la cuenta protegida por contraseña del usuario. En este estudio, el personal del proyecto de investigación administrará y será propietario de las cuentas y tendrá acceso a los datos de uso dentro de la cuenta. Dado que la cuenta no será identificable, el personal de investigación no podrá vincular estos datos de uso a familias específicas. Mantendremos datos de uso no identificables en la base de datos del proyecto de investigación. Esto incluirá datos como el tiempo dedicado a usar la habilidad, el porcentaje correcto, el progreso y la frecuencia con la que se practicó una palabra.
- 3. Usted y/o su hijo/a puede que se sientan incómodos si no están seguros de cómo responder las preguntas de las encuestas. Podrá llamarnos o enviarnos un mensaje de texto y le brindaremos asistencia.

## Beneficios para Usted y Su Hijo/a por Participar

Usted y su hijo pueden disfrutar aprendiendo nuevas palabras de vocabulario y usándolas para hablar sobre los intereses de la escuela y el hogar. Usted y su hijo pueden disfrutar de ser parte de una investigación que respalda los resultados educativos y de salud de los demás.

## Su Derecho a Retirarse del Estudio

Su participación es completamente voluntaria y privada. Aunque la escuela de su hijo/a haya compartido esta oportunidad de investigación con usted, nadie en la escuela de su hijo/a sabrá quién elige participar o no. Si decide no participar, no afectará a su hijo/a en la escuela. Si decide participar, puede dejar de participar en cualquier momento sin penalización.

### Solicite más información

Si tiene preguntas sobre la investigación en cualquier momento, o si tiene una discapacidad visual o de otro tipo y necesita este material en otro formato, llame a: Alexia Perez, Asistente de investigación (786)-559-6583, 3800 Sports Way, Springfield, OR 97477. El número TDD de ORI es 800-735-2900.

Si tiene preguntas sobre sus derechos como sujeto de investigación, llame a la Oficina para la Protección de Sujetos Humanos, Instituto de Investigación de Oregón, (541) 484-2123. El número TDD de ORI es 800-735-2900.

¿Tiene preguntas?

Hemos enviado una copia de este formulario a usted para guardar. Decir que sí desea participar en el estudio indica que usted:

- (1) ha comprendido la información proporcionada hoy,
- (2) acepta participar,

- (3) consiente a la participación de su hijo/a,
- (4) puede retirar su consentimiento en cualquier momento y dejar de participar en cualquier momento sin penalización,
- (5) puede retirar su consentimiento para la participación de su hijo/a en cualquier momento sin penalización para usted o su hijo/a,
- (6) ha recibido una copia de este formulario de consentimiento.

| ¿Desea participar en el estudio? Sí<br>¿Permite que su hijo/a participe en el estud | No<br>io? Sí No |
|---|---|
| Nombre completo (padre/madre) | Nombre de su hijo/a |
| Fecha | |

# Mi Familia STEM Estudio de Evaluación Acuerdo de Participación para Estudiantes

Te invitamos a ti y a tu familia a participar en un estudio para probar la aplicación Mi Familia STEM y la tecnología de altavoz inteligente. Mi Familia STEM es un juego de aprendizaje de palabras en español e inglés para teléfonos y altavoces inteligentes. Incluye palabras como: evidencia, variable, dimensión e hipótesis y otras palabras que ayudan a los estudiantes en la escuela.

Si decides participar, te pediremos que uses Mi Familia STEM durante aproximadamente 10 minutos, 3 veces por semana, durante 6 meses.

También te pediremos que completes algunas encuestas en línea.

Tú y tus padres recibirán un altavoz inteligente para mantener y \$200.

Tus padres ya nos han dicho que está bien que participes si quieres. No tienes que participar si no quieres.

Si decides que deseas participar ahora, puedes cambiar de opinión en cualquier momento.

| or decides que deseas participar anora, pue | ucs c |
|---------------------------------------------|-------|
| ¿Tienes preguntas? | |
| ¿Te gustaría participar en el estudio? Sí | No |
| Nombre del estudiante: | |